CLINICAL TRIAL: NCT03655275
Title: The Effects of Platelet-rich Plasma Prolotherapy on Pain Score and Frequency of Luxation in Temporomandibular Joint Subluxation A Prospective Randomized Placebo Controlled Trial
Brief Title: Effects of Platelet-rich Plasma Prolotherapy of Temporomandibular Joint Subluxation
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abdelrahman Soliman Alateyh (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Abdelrahman Soliman Alateyh, Principal Investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMJ prolotherapy
Record Dates: First submitted 2018-08-26; First posted 2018-08-31 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Temporomandibular Joint Disorders
Keywords: subluxation , platelet rich plasma (PRP), prolotherapy.
MeSH Terms: conditions — Temporomandibular Joint Disorders; Joint Dislocations

STUDY DESIGN:
Intervention Model Description: This study is randomized, placebo controlled trial.
Masking Description: This study is randomized, placebo controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group(A): PRP (Active Comparator): PRP prolotherapy injections with 2.5ml of PRP at an interval of 2 weeks. Intraticular and pericapsular
  Interventions: Biological: PRP prolotherapy
- Group (B): saline (Active Comparator): Saline prolotherapy injections with 2.5ml of saline at an interval of 2 weeks.intrarticular and pericapsular
  Interventions: Biological: Saline prolotherapy

INTERVENTIONS:
Biological: PRP prolotherapy — PRP prolotherapy By injection 2.5ml of PRP at an interval of 2 weeks.
  Arms: Group(A): PRP
Biological: Saline prolotherapy — Saline prolotherapy Injection 2.5 ml of saline at an interval of 2 weeks.
  Arms: Group (B): saline

SUMMARY:
The aim of this study is to clinically assess the efficacy of PRP prolotherapy for treatment of TMJ subluxation

DETAILED DESCRIPTION:
The effect of platelet-rich plasma prolotherapy on the pain score and frequency of luxation in temporomandibular joint subluxation. A prospective randomized placebo controlled trial

* After detailed clinical evaluation, every patient will undergo routine preoperative laboratory tests (complete blood cell count, HCV , HBV , Tomogram of TMJ examination). In cases in which special diagnostic procedures will be needed for more detailed evaluation of the patients, they will also be performed.
* All cases will undergo to withdraw 40 ml of blood from the patient's upper limb cubital vein using an 18G needle, subsequently 5 ml of citrate sodium solution is added to the sample as an anticoagulant. One milliliter of the blood sample will be sent for complete blood count.
* To prepare of high concentration PRP the blood sample will be then centrifuged for 15 minutes at 1600 rpm resulting in three layers: the lower layer made up of red blood cells, the intermediate layer is composed of white blood cells, and the upper layer is composed of plasma. The Buffy coat layer and the plasma layer will be later collected and centrifuged for another 7 minutes at 2800 rpm in order to concentrate platelets. The final product will be about 4-6 mL of PRP containing leukocytes.
* the skin surface of the preauricular area will be disinfected with Betadine surgical scrub solution. The anatomic landmarks will be located by asking the patient to open widely to allow drawing of the articular fossa and then to close lightly on the posterior teeth to draw the condyle within the glenoid fossa.
* Typically, each joint had 3 injection sites:
* The needle will be inserted at lateral margin of the glenoid fossa and 0.5 ml of the PRP will be slowly injected at the superior capsular attachment .Then needle will be directed immediately under the lateral margin of the glenoid fossa superiorly and medially toward the apex of the fossa.1ml of the PRP will be then slowly injected into the superior joint space
* The needle will be inserted at the condylar neck and 0.5 ml of the PRP will be injected at the inferior capsular attachment. Then needle will be directed superficial to the TMJ capsule, 0.5 ml of the PRP will be deposited as needle will be withdrawn.
* patients in the placebo group received injections of placebo (saline) using the same volume on the same schedule.
* Post operative care and instructions:
* Bleeding from the injection sites will be generally minimal and could be controlled with direct pressure on the injection site for a few seconds.
* All patients will be advised to take "paracetamol", one tablet when needed and to stop the use of other pain and anti-inflammatory drugs during the treatment phase.
* Each patient will be instructed to receive soft diet only for two weeks in order to decrease the effort upon TMJ .

ELIGIBILITY:
Inclusion Criteria:

1. Patients who had TMJ subluxation for at least six months.
2. Age ≥ 18 years
3. Willingness of the patient to receive relative painful injections and to follow instructions.

Exclusion Criteria:

* 1. Patients with dystonia 2. Drug induced TMJ hypermobility 3. Medical conditions that could significantly interfere with treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2018-08-24 (Estimated); Primary Completion 2018-09-30 (Estimated); Study Completion 2019-05-30 (Estimated)

PRIMARY OUTCOMES:
Patients' subjective pain experience | up to 40 weeks
  visual anlogue scale (VAS) from 0 - 10

SECONDARY OUTCOMES:
Frequency of luxation | up to 40 weeks
  The number of luxation/day
Maximum mouth opening | up to 40 weeks
  ruler per mm from 0 - 70
Joint sounds | up to 40 weeks
  preauricular palpation

CONTACTS AND LOCATIONS:
Overall Officials: Hamida R Hassanien, phd, Study Director — Cairo University
Locations (1):
- Faculty of Oral and Dental Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Group A : each joint will receive 2 session of intrarticular and pericapsular injections with 2.5ml of PRP at interval of 2 weeks.
  • Group B : : each joint will receive 2 session of intrarticular and pericapsular injections with 2.5ml of PRP at interval of 2 weeks.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: few months to year
Access Criteria: The effects of platelet-rich plasma prolotherapy on pain score and frequency of luxation in temporomandibular joint subluxation A prospective randomized placebo controlled trial

REFERENCES:
- [Background] Middleton KK, Barro V, Muller B, Terada S, Fu FH. Evaluation of the effects of platelet-rich plasma (PRP) therapy involved in the healing of sports-related soft tissue injuries. Iowa Orthop J. 2012;32:150-63. PMID 23576936
- [Background] Pihut M, Szuta M, Ferendiuk E, Zenczak-Wieckiewicz D. Evaluation of pain regression in patients with temporomandibular dysfunction treated by intra-articular platelet-rich plasma injections: a preliminary report. Biomed Res Int. 2014;2014:132369. doi: 10.1155/2014/132369. Epub 2014 Aug 3. PMID 25157351
- [Background] Jureidini J. Is there a role for placebo analgesia? N Z Med J. 2003 Aug 8;116(1179):U541. No abstract available. PMID 14513087
- [Background] Yelland MJ, Glasziou PP, Bogduk N, Schluter PJ, McKernon M. Prolotherapy injections, saline injections, and exercises for chronic low-back pain: a randomized trial. Spine (Phila Pa 1976). 2004 Jan 1;29(1):9-16; discussion 16. doi: 10.1097/01.BRS.0000105529.07222.5B. PMID 14699269